CLINICAL TRIAL: NCT01157650
Title: Treatment of Fistulous Crohn's Disease by Implant of Autologous Mesenchymal Stem Cells Derived From Adipose Tissue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/CROH; 2009-009880-71 (EudraCT Number)
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Crohn Disease
Keywords: Fistulizing Crohn's disease; stem cells implant
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous mesenchymal stem cells (Experimental): Fistulizing Crohn's disease
  Interventions: Other: Autologous mesenchymal stem cells

INTERVENTIONS:
Other: Autologous mesenchymal stem cells — The trial is divided in three phases:
  I. - Selection: Patients evaluation for study eligibility will take place within two weeks after Informed Consent signature.
  II.- Treatment phase includes:
  1. Liposuction procedure to obtain adipose tissue.
  2. Processing and production of Autologous Mesenchymal Stem Cells from adipose tissue (ASCs)
  3. ASCs implant
  III.- Follow up: Study visits post-implant will take place at the 1st week (+/- 3 days), 4th week (+/- 3 days), 8th week (+/- 7 days), 12nd week (+/- 7 days), 24th week (+/- 7 days), and 1 year (+/- 7 days) after implant.
  Other Names: Implant of ASCs.

SUMMARY:
Primary outcome measure:

Evaluation of viability, security and tolerance of the adipose-derived mesenchymal stem cells implant (ASCs) in fistulizing Crohn's disease patients, collecting the reactions and adverse events occurred during the study.

Secondary outcome measures:

1. Evaluating the Adipose-derived mesenchymal stem cells therapeutic effect, in particular:

   * Fistulas healing efficiency
   * Changes in quality of life in patients treated
   * Changes of systemic Crohn's disease after implant
   * Relapse rate monitored among patients who achieved Adipose-derived mesenchymal Stem Cells treatment success.
2. Achieving the biological characterization of the cell product used and its correlation with the therapeutic effect measured with:

   * Phenotype study
   * Suppressor capacity study.
   * Citoquines production analysis

DETAILED DESCRIPTION:
The aim of this study is to evaluate the role of Autologous Mesechymal Stem Cells derived from adipose tissue in the treatment of fistulous Crohn disease.

15 Crohn's disease patients with one or more enterocutaneous, recto-vaginal or complex perianal fistula, will be included.

The trial is divided in three phases:

I. - Selection: Patients evaluation for study eligibility will take place within two weeks after Informed Consent signature.

Fistulous disease will be evaluated by MRI for perianal and rectovaginal fistulas, and by CT scan in the case of enterocutaneous fistula.

Previous laboratory test and radiological studies are valid for evaluation if they were obtained within two and six months, respectively, prior to this evaluation, and in the absence of clinical changes.

II.- Treatment phase includes:

1. Liposuction procedure to obtain adipose tissue.
2. Processing and production of Autologous Mesenchymal Stem Cells from adipose tissue (ASCs)
3. ASCs implant

III.- Follow up: Study visits post-implant will take place at the 1st week (+/- 3 days), 4th week (+/- 3 days), 8th week (+/- 7 days), 12nd week (+/- 7 days), 24th week (+/- 7 days), and 1 year (+/- 7 days) after implant.

ELIGIBILITY:
Inclusion Criteria:

1. Fistulizing Crohn´s disease patients with 1 or more enterocutaneous fistulas, recto-vaginal fistula or complex perianal fistula. The complex perianal fistula is defined as a fistula presenting one of these conditions:

   * Trans-sphincteric, supra-sphincteric or extra-sphincteric tract, determined with:
   * Clinical criteria: No palpation of the tract and surgical exploration
   * Radiological criteria: Nucleal Magnetic Resonance (NMR)or Echoendoscopy
   * Multiple fistulas
   * "Horseshoe" fistula
   * Any fistula with fecal incontinence associated
   * Any fistula with a risk of fecal incontinence as a result of:
   * previous anal fistula surgery or other perianal pathology (hemorrhoids, fissures), that involves lesions or muscular complications.
   * Obstetric or iatrogenic sphincter lesions
2. Patients with Crohn Disease (CD) at screening and been diagnosed within 12 months before acceptance of clinical, endoscopical, anatomopathological and/or radiological criteria and have a non-active CD.(Crohn´s Disease Activity Index (CDAI)≤ 200)
3. > 18 Years and both genders eligible.
4. Negative pregnancy test In female fertile subjects
5. Patient must voluntary sign the informed consent before performance of any study-related procedure not part of normal medical care.
6. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements

Exclusion Criteria:

1. Patients with a highly active CD, i.e., if they meet any of the following criteria:

   * Presence of severe proctitis (prominent friability, spontaneous bleeding, multiple erosions, deep ulcers) or dominant active luminal disease that requires immediate treatment, revealed by rectosigmoidoscopy
   * CDAI ≥201
2. Presence of abscess or other collections not drained (revealed by basal radiologic study).
3. Presence of setons drainage, unless they are removed before treatment beginning.
4. Rectal and/ or anal stenosis revealed with rectoscopy or EBA.
5. Patients needs surgery in the perianal region for other reasons than fistulas at inclusion or within 26 weeks after treatment administration.
6. Patients who have received infliximab or any other anti-TNF agent within 8 weeks before the cell treatment administration.
7. Patients who have received tacrolimus or cyclosporine within 4 weeks before cell treatment.
8. Patients with a history of alcohol or other addictive substances abuse within 6 months before inclusion.
9. Severe uncontrolled diseases (chronic renal failure, cardio, pulmonary,…).
10. Any type of medical or psychiatric disease which are considered as exclusion criteria, in the investigator's opinion.
11. Patients with diagnosis of malignant neoplasia, except basal cell or epidermoid carcinoma of the skin or previous history of malignant tumours, except those that have no evidence of relapse for at least 5 years.
12. Subjects with congenital or acquired immunodeficiency.
13. Positive serology for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV).
14. Patient had major surgery or serious traumatism within 6 weeks before enrolment.
15. Pregnant or breast-feeding women.
16. Physical or psychical impossibility of following the protocol requirements
17. Patients who are receiving or received other investigational drugs within 30 days prior to basal visit.
18. Impossibility of doing an radiological exploration (reaction to contrast material, pacemakers, claustrophobia,…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Security and tolerance | 3 years
  Evaluation of viability, security and tolerance of the adipose-derived mesenchymal stem cells implant (ASCs) in fistulizing Chron's disease patients, collecting the reactions and adverse events occurred during the study

SECONDARY OUTCOMES:
therapeutic effect | 3 years
  1. Evaluting the ASCs therapeutic effect, in particular:
     * Fistulas healing efficiency
     * Changes in quality of life in patients treated
     * Changes of systemic Crohn's disease after implant
     * Relapse rate monitored among patients who achieved ASCs treatment success.
  2. Achieving the biological characterization of the cell product used and its correlation with the therapeutic effect measured with:
     * Phenotype study
     * Suppressor capacity study.
     * Citoquines production analysis

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Prosper, MD, PhD, Study Director — Clinica Universidad de Navarra
Locations (3):
- Spain (3):
  - Clínica Universitaria de Navarra, Pamplona, Pamplona
  - Hospital Provincial de Navarra, Pamplona, Pamplona
  - Hospital Virgen del Camino, Pamplona, Pamplona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nivatvongs S, Gordon PH. Crohn's Disease. In: Gordon PH, Nivatvongs S, editors. Principles and practice of surgery for the colon rectum and anus Third ed. New York: Informa Healthcare; 2007. p. 819-908.
- [Background] Brullet E, Bonfill X, Urrutia G, Ruiz Ochoa V, Cueto M, Clofent J, Martinez Salmeron JF, Riera J, Obrador A. [Epidemiological study on the incidence of inflammatory bowel disease in 4 Spanish areas. Spanish Group on the Epidemiological Study of Inflammatory Bowel Disease]. Med Clin (Barc). 1998 May 16;110(17):651-6. Spanish. PMID 9656209
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Arin Letamendia A, Borda Celaya F, Burusco Paternain MJ, Prieto Martinez C, Martinez Echeverria A, Elizalde Apestegui I, Laiglesia Izquierdo M, Macias Mendizabal E, Tamburri Moso P, Sanchez Valverde F. [High incidence rates of inflammatory bowel disease in Navarra (Spain). Results of a prospective, population-based study]. Gastroenterol Hepatol. 2008 Mar;31(3):111-6. doi: 10.1157/13116497. Spanish. PMID 18341841
- [Background] Lapidus A, Bernell O, Hellers G, Lofberg R. Clinical course of colorectal Crohn's disease: a 35-year follow-up study of 507 patients. Gastroenterology. 1998 Jun;114(6):1151-60. doi: 10.1016/s0016-5085(98)70420-2. PMID 9609751
- [Background] Parsi MA, Lashner BA, Achkar JP, Connor JT, Brzezinski A. Type of fistula determines response to infliximab in patients with fistulous Crohn's disease. Am J Gastroenterol. 2004 Mar;99(3):445-9. doi: 10.1111/j.1572-0241.2004.04083.x. PMID 15056083
- [Background] Michelassi F, Stella M, Balestracci T, Giuliante F, Marogna P, Block GE. Incidence, diagnosis, and treatment of enteric and colorectal fistulae in patients with Crohn's disease. Ann Surg. 1993 Nov;218(5):660-6. doi: 10.1097/00000658-199321850-00012. PMID 8239781
- [Background] Gardiner KR, Dasari BV. Operative management of small bowel Crohn's disease. Surg Clin North Am. 2007 Jun;87(3):587-610. doi: 10.1016/j.suc.2007.03.011. PMID 17560414
- [Background] Hyder SA, Travis SP, Jewell DP, McC Mortensen NJ, George BD. Fistulating anal Crohn's disease: results of combined surgical and infliximab treatment. Dis Colon Rectum. 2006 Dec;49(12):1837-41. doi: 10.1007/s10350-006-0656-5. PMID 17041753
- [Background] Gelbmann CM, Rogler G, Gross V, Gierend M, Bregenzer N, Andus T, Scholmerich J. Prior bowel resections, perianal disease, and a high initial Crohn's disease activity index are associated with corticosteroid resistance in active Crohn's disease. Am J Gastroenterol. 2002 Jun;97(6):1438-45. doi: 10.1111/j.1572-0241.2002.05685.x. PMID 12094862
- [Background] Pearson DC, May GR, Fick GH, Sutherland LR. Azathioprine and 6-mercaptopurine in Crohn disease. A meta-analysis. Ann Intern Med. 1995 Jul 15;123(2):132-42. doi: 10.7326/0003-4819-123-2-199507150-00009. PMID 7778826
- [Background] Lecomte T, Contou JF, Beaugerie L, Carbonnel F, Cattan S, Gendre JP, Cosnes J. Predictive factors of response of perianal Crohn's disease to azathioprine or 6-mercaptopurine. Dis Colon Rectum. 2003 Nov;46(11):1469-75. doi: 10.1007/s10350-004-6795-7. PMID 14605564
- [Background] Sandborn WJ, Present DH, Isaacs KL, Wolf DC, Greenberg E, Hanauer SB, Feagan BG, Mayer L, Johnson T, Galanko J, Martin C, Sandler RS. Tacrolimus for the treatment of fistulas in patients with Crohn's disease: a randomized, placebo-controlled trial. Gastroenterology. 2003 Aug;125(2):380-8. doi: 10.1016/s0016-5085(03)00877-1. PMID 12891539
- [Background] Present DH, Lichtiger S. Efficacy of cyclosporine in treatment of fistula of Crohn's disease. Dig Dis Sci. 1994 Feb;39(2):374-80. doi: 10.1007/BF02090211. PMID 8313821
- [Background] Hanauer SB, Smith MB. Rapid closure of Crohn's disease fistulas with continuous intravenous cyclosporin A. Am J Gastroenterol. 1993 May;88(5):646-9. PMID 8480725
- [Background] Present DH, Rutgeerts P, Targan S, Hanauer SB, Mayer L, van Hogezand RA, Podolsky DK, Sands BE, Braakman T, DeWoody KL, Schaible TF, van Deventer SJ. Infliximab for the treatment of fistulas in patients with Crohn's disease. N Engl J Med. 1999 May 6;340(18):1398-405. doi: 10.1056/NEJM199905063401804. PMID 10228190
- [Background] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485
- [Background] Poritz LS, Rowe WA, Koltun WA. Remicade does not abolish the need for surgery in fistulizing Crohn's disease. Dis Colon Rectum. 2002 Jun;45(6):771-5. doi: 10.1007/s10350-004-6296-8. PMID 12072629
- [Background] García-Olmo D, Trébol J, et al. Treatment of digestiva fistula using Adipose-derived Stem Cells. In: García-Olmo D, García-Verdugo JM, Alemany J, Gutierrez-Fuentes JA, editors. Cell Therapy. Madrid: McGraw-Hill. Interamericana; 2008. p. 289-307.
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Result] Thoreson R, Cullen JJ. Pathophysiology of inflammatory bowel disease: an overview. Surg Clin North Am. 2007 Jun;87(3):575-85. doi: 10.1016/j.suc.2007.03.001. PMID 17560413